CLINICAL TRIAL: NCT02316015
Title: Protein-energy Enriched Milk for Infants With Bronchiolitis
Acronym: PEMIB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Koen Huysentruyt, Dr., Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: B.U.N. 143201422489
Record Dates: First submitted 2014-12-05; First posted 2014-12-12 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Bronchiolitis
Keywords: Child, Hospitalized; Nutritional status
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Children in the intervention group will receive a protein-energy enriched milk (Infatrini®, or in the case of children on a partial or fully hydrolized milk Infatrini Peptisorb®). The volume of milk offered will be the same quantity as they usually drink at home (within the limits of 120-170 ml/kg/day). The intervention will be carried out during the first 7 days of hospitalisation, or until the day of discharge (if hospitalized for less than 7 days).
  Interventions: Dietary Supplement: Infatrini® or Infatrini Peptisorb®
- Control group (No Intervention): Children in the control group will receive their regular milk. The volume of milk offered will be the same quantity as they usually drink at home (within the limits of 120-170 ml/kg/day).

INTERVENTIONS:
Dietary Supplement: Infatrini® or Infatrini Peptisorb®
  Arms: Intervention group

SUMMARY:
The aim of this study is to investigate if a standardized nutritional intervention with a protein and energy enriched milk could help overcome the catabolic state in children hospitalized with a bronchiolitis and thus creating a better nutritional state during hospitalization and at outpatient follow-up.

The investigators also want to assess the clinical repercussion on the number of hospitalization days, the duration of oxygen support and the quality of life at ouptatient follow-up.

DETAILED DESCRIPTION:
In this study, the investigators aim to assess the effect protein-energy enriched milk to reverse the catabolic state (weight loss, change in mid-upper arm circumference and tricpes skin fold) on the short term and failure to thrive (degree of weight recovery, change in arm circumference) one week after discharge in infants with moderate to severe bronchiolitis. The secondary short term aims are to investigate the effect on the length of hospital stay, days of oxygen support and the rate of antibiotic use. Secondary long term outcomes are the re-admission rate, the persistence of wheezing and the number of work days missed by the parents.

The investigators hypothesize that in those children who received a protein-energy enriched milk during hospitalization the catabolic state will be reversed more quickly by the intervention and will need less hospitalisation days, less oxygen support, less antibiotic use, less re-admission rate, less persistent wheezing and less work days missed by the parents. The investigators also hypothesize that the effects of the nutritional intervention on the proposed outcome parameters will be greater in children screened at high nutritional risk.

ELIGIBILITY:
Inclusion Criteria:

* All children hospitalized at the paediatric wards of UZ Brussel with the diagnosis of moderate to severe bronchiolitis
* Not meeting their normal oral intake are eligible for inclusion between the beginning of December and the end of February 2014
* Bronchiolitis will be defined as a constellation of clinical symptoms and signs that typically begin with rhinitis and cough, and may progress to tachypnea, wheezing, rales, use of accessory muscles and/or nasal flaring

Exclusion Criteria:

* Children admitted to the paediatric intensive care unit
* Children in whom it is unsafe to place a nasogastric tube (e.g. severe mucositis, platelet count <50.000/µl)
* Children unwilling or unable to participate
* Children that are breast fed
* Children over the age of 12 months
* Children with an underlying malabsorption disease

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Evolution of nutritional status during hospitalization | Hospital stay (mean 5 days)
  The change in followong parameters will be assessed:
  * Change in weight for age z-score
  * Change in mid upper arm circumference z-score
  * Change in triceps skin fold (mm)

SECONDARY OUTCOMES:
Evolution of nutritional status at outpatient follow-up | 1 week after discharge
  - Change in WFA z-score, weight for height z-score, MUAC z-score and TSF (mm)

OTHER OUTCOMES:
The Quality of life at outpatient follow-up | 1 week after discharge
  The ITQOL-SF47 questionnaire will be used to assess quality of life
Duration of hospital stay | Hospital stay (mean 5 days)
  Number of days of hospitalization
Time of oxygen support | Hospital stay (mean 5 days)
  Number of hours of oxygen support during hospital stay
Rate of antibiotic use | Hospital stay (mean 5 days)
  Number of children in which antibiotics is commenced during their hospitalization
Re-admission rate | 1 week after discharge
  Number of children that are re-admitted to the hospital in the first two months after discharge
Persistence of wheezing | 1 week after discharge
  This will be assessed using the respiratory distress assessment instrument (Langley et al., 2005)

CONTACTS AND LOCATIONS:
Overall Officials: Yvan Vandenplas, MD, PhD, Principal Investigator — UZBrussel
Locations (1):
- UZ Brussel, Jette, Belgium